CLINICAL TRIAL: NCT03928548
Title: Malnutrition Clinical Characteristics Validation and Staffing Optimization Study
Brief Title: Malnutrition Clinical Characteristics Validation and Staffing Optimization Study (MCC Study)
Status: Completed | Type: Observational
Sponsor: Academy of Nutrition and Dietetics (Other)
Responsible Party: Sponsor
Other Study IDs: 18-594
Record Dates: First submitted 2019-04-10; First posted 2019-04-26 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Risk Malnutrition: Participants who are determined to be at low risk for malnutrition based on the Malnutrition Screening Tool (adults) or the STRONGkids (pediatrics).
- High Risk Malnutrition: Participants who are determined to be at high risk for malnutrition based on the Malnutrition Screening Tool (adults) or the STRONGkids (pediatrics).

SUMMARY:
The purpose of this study is to establish the validity of the adult and pediatric Malnutrition Clinical Characteristics (MCC). In addition, this project will: examine the relationship between the MCC and an objective measure of body composition; and establish the relationship between in-patient Registered Dietitian Nutritionist (RDN) care and medical outcomes for all in-patients requiring nutrition care, and specifically for malnourished patients. Sixty pediatric and 60 adult in-patient acute care facilities will participate in this research study. The total number of participants enrolled across the 120 facilities will be between 2400-9600.

The aims of the study include:

1. Assess the interrater reliability of the MCC.
2. Determine the predictive validity of the adult and pediatric MCC relative to a portfolio of patient medical outcomes.
3. Determine the relationship between the adult and pediatric MCC and body composition measurements conducted via bioelectrical impedance analysis (BIA) in a subset of patients.
4. Identify the utility of BIA for body composition analysis in clinical settings.
5. Estimate the level of RDN care necessary to improve patient outcomes within the portfolio of outcomes. Specifically: quantify the dose (minutes of care and frequency of encounters) of RDN care that is associated with improved medical outcomes in patients already identified as requiring nutrition care, after adjusting for disease severity and other potential confounders.
6. Identify the additional level of RDN care necessary to improve the medical outcomes in patients who have been identified as malnourished using the MCC.

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric acute care patients at participating facility
* Newly identified as needing in-patient nutrition care through current facility policy
* Receive initial nutrition care one day before study enrollment day
* Patient is over one month of age, including infants, children, teenagers and adult patients who are intubated and/or sedated
* Patient, parent, legal guardian or legally authorized representative provide informed consent; children 7 and older provide assent
* Patient and/or parent, legal guardian or legally authorized representative are fluent in English or Spanish

Exclusion Criteria:

* Received nutrition care previously during current admission
* Pregnant women
* Prisoners
* Infants currently in the neonatal intensive care unit (NICU) with a diagnosis of prematurity
* Neonates of uncertain viability or non-viable neonates
* Patients receiving palliative/hospice care
* Patient admitted for long-term acute care (LTAC)

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients (according to the inclusion and exclusion criteria seen below) who are admitted to the participating hospitals in the United States.
Sampling Method: Probability Sample
Enrollment: 887 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Length of stay | 90 Days
  Number of days a participant is in-patient at an acute care hospital (discharge date - admission date) as measured by the existing medical record
Post-discharge readmissions | 90 Days
  Number of times a participant is readmitted to the hospital after the initial discharge as measured by the existing medical record
Post discharge emergency department (ED) visits | 90 Days
  Number of times a participant visits the ED after the initial discharge as measured by the existing medical record
Mortality | 90 Days
  Participant death as measured by the existing medical record

CONTACTS AND LOCATIONS:
Overall Officials: Alison Steiber, PhD, RDN, Principal Investigator — Academy of Nutrition and Dietetics
Locations (2):
- United States (2):
  - AdventHealth, Daytona Beach, Florida
  - The Children's Mercy Hospital, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez EY, Lamers-Johnson E, Long JM, McCabe G, Ma X, Woodcock L, Bliss C, Abram JK, Steiber AL. Predictive validity of the Academy of Nutrition and Dietetics/American Society for Parenteral and Enteral Nutrition indicators to diagnose malnutrition tool in hospitalized adults: a cohort study. Am J Clin Nutr. 2024 Mar;119(3):779-787. doi: 10.1016/j.ajcnut.2023.12.012. Epub 2024 Feb 12. PMID 38432715
- [Derived] Jimenez EY, Lamers-Johnson E, Long JM, Mordarski BA, Ma X, Steiber A. Completion of a Nutrition-Focused Physical Exam with hospitalized adults and pediatric patients: Secondary analysis of a prospective cohort study. Nutr Clin Pract. 2024 Aug;39(4):888-902. doi: 10.1002/ncp.11137. Epub 2024 Feb 19. PMID 38372592
- [Derived] Lamers-Johnson E, Will VK, Long JM, Woodcock L, Kelley K, Steiber AL, Jimenez EY. Factors Associated with IRB Review Time in a Non-Federally Funded Study Using an sIRB of Record. Ethics Hum Res. 2023 Jul-Aug;45(4):16-29. doi: 10.1002/eahr.500173. PMID 37368522
- [Derived] Jimenez EY, Long JM, Lamers-Johnson E, Woodcock L, Bliss C, Lee J, Scott Parrott J, Hand RK, Kelley K, Abram JK, Steiber A. Academy of Nutrition and Dietetics Nutrition Research Network: Rationale and Protocol for a Study to Validate the Academy of Nutrition and Dietetics/American Society for Parenteral and Enteral Nutrition Consensus-Derived Diagnostic Indicators For Adult And Pediatric Malnutrition and to Determine Optimal Registered Dietitian Nutritionist Staffing in Acute Care Hospital Settings. J Acad Nutr Diet. 2022 Mar;122(3):630-639. doi: 10.1016/j.jand.2021.03.017. Epub 2021 May 4. PMID 33962901